CLINICAL TRIAL: NCT00063336
Title: Treatment Response to Rehabilitation in Schizophrenia
Brief Title: Treatment Response to Rehabilitation in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Matthew M. Kurtz, PhD, Schizophrenia Rehabilitation Program, Institutes of Living
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: R03MH065377 (NIH); R03MH065377 (NIH); DSIR AT-SP
Record Dates: First submitted 2003-06-25; First posted 2003-06-27 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2009-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Remediation

ARMS (2):
- 1 (Experimental): Participants will receive cognitive remediation treatment.
  Interventions: Behavioral: Cognitive Remediation
- 2 (Experimental): Participants will receive computer-skills training.
  Interventions: Behavioral: Computer-skills training

INTERVENTIONS:
Behavioral: Cognitive Remediation — A computerized cognitive rehabilitation treatment with day-program activities
  Arms: 1
Behavioral: Computer-skills training — A computerized cognitive rehabilitation treatment with day-program activities
  Arms: 2

SUMMARY:
This study will examine the ways in which schizophrenia-related symptoms affect response to a rehabilitation program for people with schizophrenia.

DETAILED DESCRIPTION:
Patients with schizophrenia often suffer neurocognitive impairment and psychosocial and vocational difficulties. This study will help identify those patients most likely to benefit from existing behavioral treatments and provide clues for how to modify treatments for those who do not benefit.

Two studies will be conducted. The first will investigate the relationship of symptoms and neurocognitive variables at study entry to psychosocial and vocational status 2 years later. The second study will investigate the relationship of symptoms and neurocognitive variables at study entry to treatment response in patients assigned to either a cognitive remediation track or a computer skills track as part of their rehabilitation treatment.

Both the cognitive remediation and computer skills training programs will last 4 to 6 months. Participants will be assessed pre- and post-treatment. Neuropsychological, psychosocial and vocational status will be measured.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for schizophrenia or schizoaffective disorder
* In need of intensive outpatient care
* Treatment with atypical antipsychotic medication for a minimum of 6 months prior to study entry

Exclusion Criteria:

* Auditory or visual impairment
* Mental retardation (IQ less than 70)
* Traumatic brain injury with loss of consciousness
* Presence or history of any neurological illness that may affect brain physiology
* Lack of proficiency in English
* Concurrent substance abuse and/or dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2001-12; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Neuropsychological test battery, including measures of visual, verbal memory, and problem-solving abilities | Measured pre- and post-treatment
Schizophrenia symptoms | Measured pre- and post-treament
UCSD Performance-Based Skills Assessment | Measured pre- and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M. Kurtz, PhD, Principal Investigator — Schizophrenia Rehabilitation Program, Institutes of Living
Locations (1):
- Schizophrenia Rehabilitation Program, Institutes of Living, Hartford, Connecticut, United States